CLINICAL TRIAL: NCT01006967
Title: Randomized ActiveStep Comparative Effectiveness Trial
Brief Title: ActiveStep Comparative Effectiveness Trial
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jon D. Lurie (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jon D. Lurie, Professor of Medicine (General Internal Medicine), Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AHRQ R18 HS18459
Record Dates: First submitted 2009-10-27; First posted 2009-11-03 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Gait Disorders
Keywords: balance; accidental falls; physical therapy; ActiveStep; older adults
MeSH Terms: conditions — Mobility Limitation | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ActiveStep (Active Comparator): Subjects will use the ActiveStep treadmill as part of their physical therapy program for balance
  Interventions: Device: ActiveStep Treadmill
- Standard physical therapy (Active Comparator): Subjects will receive a standard physical therapy program for gait and balance.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: ActiveStep Treadmill — The ActiveStep treadmill is a device that trains patients to effectively react to simulated slips and trips while the patient is safely held in a harness.
  Arms: ActiveStep
Other: Physical Therapy — Standard program of physical therapy for gait and balance
  Arms: Standard physical therapy

SUMMARY:
The investigators are conducting a multi-center randomized prospective trial comparing a standard physical therapy gait and balance program with a gait and balance program that includes the ActiveStep™ treadmill.

Subjects will be randomized to either have the ActiveStep™ as part of their therapy or to have their therapy without it. Data will be gathered from session notes, medical records and short interviews with the subjects at baseline and every 3 months over the telephone for the duration of the study.

DETAILED DESCRIPTION:
Falls are the leading cause of fatal and non-fatal injuries in the elderly. Each year an estimated 1/3 of older adults fall, and the likelihood of falling increases substantially with advancing age.2 In 2005, 15,802 elderly patients (> 65 years of age) died as the result of fall-related injuries. According to the 2006 Behavioral Risk Factor Surveillance System (BRFSS) survey, 5.8 million persons aged 65 or older fell at least once during a 3 month period, which represents nearly 16 percent of the elderly population; furthermore, nearly a third of those who fell (1.8 million) sustained some form of injury that resulted in either a doctor's visit or restricted activity for at least 1 day. Falls thus represent a major cause of functional limitation and disability in the elderly. In 2000, the direct medical costs for fall-related injuries was estimated to be $19 billion. Our primary objective is to perform a multi-center, randomized clinical trial to evaluate the comparative effectiveness of a perturbation-based dynamic stability intervention (using the ActiveStep® training system) compared to a traditional physical therapy program in reducing the incidence and severity of falls in a geriatric population.

Modifiable risk factors for falls include muscle weakness, gait and balance problems, poor vision, use of psychoactive medications, and home hazards. Most effective fall-prevention interventions focus on exercise, either alone or as part of a multi-faceted program including medication management, vision correction and home modifications. One Tai Chi based program reduced the risk of falls by 55% in a randomized trial. While exercise programs appear to have efficacy in reducing fall risk, the type, frequency and duration of exercise that is adequate to significantly reduce the risk of falls remain unclear.

External perturbations such as tripping are a major contributor to falls, and trip-related falls account for as many as 20% of all hip fractures.

The ActiveStep® fall prevention training program was developed with NIH funding and consists of a series of increasingly challenging postural disturbances using a microprocessor controlled servo motor that drives a treadmill belt at defined acceleration, velocity, and distance profiles. Initial biomechanical testing of the ActiveStep® training program showed significant improvement in trunk kinematics during a single training session. The ActiveStep® training program is currently available and billable under Medicare reimbursement codes; however, there is a lack clinical data showing that it can reduce falls during patients' routine activities better than standard physical therapy interventions.

The Specific Aims are to:

1. To conduct a prospective, multi-center, pragmatic, randomized comparative effectiveness trial comparing a standard physical therapy gait and balance program with a perturbation-based dynamic stability intervention using the ActiveStep® training system. The main outcome measures were the number of subjects who reported a fall and the number who reported an injurious fall during the follow-up periods. Secondary measures included the subjects' self-reported balance confidence using the Activities-specific Balance Confidence (ABC) scale.
2. To assess the longevity of any improvement with the two types of fall prevention programs by assessing falls every three months out to at least one year. The data on time to first fall will allow insight into the potential need for and timing of "retraining" for fall prevention.
3. To evaluate for underlying patient characteristics that may predict successful prevention of falls in both treatment groups and thus help with determining appropriate selection of patients into different types of fall prevention programs.

Men and women 65 years or older who are referred for fall prevention physical therapy intervention will be eligible for the Randomized ActiveStep® Comparative Effectiveness Trial (RACE Trial). Patients will either have had a prior fall or score as a fall risk on at least one of the balance assessment measure as described below. Following education about the study and participation in the informed consent process, patients who agree to participate will be randomly assigned to either standard physical therapy gait-and-balance training (PT) or to PT+ActiveStep® in a one-to-one ratio. The study will not be blinded as there is no adequate sham-control for the ActiveStep® training; however, allocation concealment will be ensured until after patients are enrolled. The final planned target enrollment will be 550 subjects.

At the time of enrollment, all participants will undergo a fall risk assessment. This will include several standard instruments including: the Timed Up & Go Test (TUG); 42 the Dynamic Gait Index (DGI); 43 and the Berg Balance Measure. 44 In addition we will administer the Activities-specific Balance Confidence (ABC) scale, a questionnaire that assesses the level of self-confidence the patient has in their balance during 16 specific activities. 45 This scale does not assess fall risk per se but does assess fear of falling that can have a significant impact on patients' activity levels and quality of life.

The treatment protocol for the PT cohort will consist of current standard gait / balance training physical therapy as described below. The PT+ActiveStep® will receive standard PT training but with the inclusion of a number of 15 minute sessions on the ActiveStep® simulator. The content of the standard PT in the ActiveStep® group will be adjusted such that the total number of rehabilitation visits and amount of rehabilitation time will be the same for both groups, taking into account the maximum number of allowable visits for reimbursement. Thus, the ActiveStep® will substitute for some portion of the standard PT intervention.

Following the treatment phase, study subjects will be contacted by telephone every 3 months for the duration of the study for a brief interview regarding their history of falling and any significant changes in medical condition. The primary question of interest is the potential difference between treatment groups in the ability to reduce the occurrence of injurious falls subsequent to treatment. This question will be evaluated in two different ways. First, the proportion of subjects in each group experiencing a fall or an injurious fall at each timepoint will be compared; this will allow direct comparison to the three month outcomes of the pilot trial. Second, survival analysis will be used to evaluate for group differences in the likelihood of a post-treatment injurious fall over the follow-up period. In this approach the survival analysis will predict time to first injurious fall. Both of these analyses will include relevant baseline patient characteristics and pre- to post-treatment changes in functioning in an attempt to identify factors or constellations of factors that might predict subsequent fall risk. Secondary analyses will look for the occurrence of any falls using negative binomial regression to allow for the occurrence of multiple falls per subject over time.

Comorbid factors gathered as part of the follow-up process, such as medication use and co-morbidity status, will be evaluated across treatment groups using simple maximum likelihood chi-square tests. Additionally, changes in the TUG, Berg, DGI, or ABC scales before and after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over
* Referred to physical therapy for balance training

Exclusion Criteria:

* Age < 65
* Unable to use treadmill
* Severe vertigo
* Not a candidate for gait/balance PT
* Not competent to consent to research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 506 (Actual)
Dates: Start 2009-11; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Lurie, M.D., M.S., Principal Investigator — Dartmouth College
Locations (8):
- United States (8):
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Spaulding Rehabilitation Hospital, Salem, Massachusetts
  - Concord Hospital Rehabilitation Services, Epsom, New Hampshire
  - Cheshire Medical Center - Farnum Rehabilitation Center, Keene, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Elliot Hospital, Manchester, New Hampshire
  - South Shore Neurological Associates, Patchogue, New York
  - White River Junction Veterans Administration Medical Center, White River Junction, Vermont

REFERENCES:
- [Derived] Lurie JD, Zagaria AB, Ellis L, Pidgeon D, Gill-Body KM, Burke C, Armbrust K, Cass S, Spratt KF, McDonough CM. Surface Perturbation Training to Prevent Falls in Older Adults: A Highly Pragmatic, Randomized Controlled Trial. Phys Ther. 2020 Jul 19;100(7):1153-1162. doi: 10.1093/ptj/pzaa023. PMID 31998949
- [Derived] Lurie JD, Zagaria AB, Pidgeon DM, Forman JL, Spratt KF. Pilot comparative effectiveness study of surface perturbation treadmill training to prevent falls in older adults. BMC Geriatr. 2013 May 16;13:49. doi: 10.1186/1471-2318-13-49. PMID 23678970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ActiveStep | Standard Physical Therapy
Started | 253 | 253
Received Treatment | 245 | 245
3 Month Follow-up | 212 | 210
Completed | 187 | 190
Not Completed | 66 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ActiveStep | Standard Physical Therapy | Total
Number analyzed (Participants) | 253 | 253 | 506
Age, Continuous [Mean (Full Range); unit: years] | 78 [65 to 96] | 78 [65 to 95] | 78 [65 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 119 | 238
  Male | 134 | 134 | 268
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fall in past 3 months [Count of Participants; unit: Participants] | 136 | 130 | 266
Fall in Past Year [Count of Participants; unit: Participants] | 179 | 169 | 348

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Fall
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | ActiveStep | Standard Physical Therapy
Number analyzed (Participants) | 212 | 210
Participants | 60 | 77

2. Primary Outcome: Number of Subjects Reporting a Fall-related Injury
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | ActiveStep | Standard Physical Therapy
Number analyzed (Participants) | 212 | 210
Participants | 12 | 28

3. Secondary Outcome: Change in Timed Up and Go From Baseline
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ActiveStep | Standard Treatment
Number analyzed (Participants) | 149 | 153
seconds | -1.96 (318) | -2.18 (3.86)

4. Secondary Outcome: Change in Berg Balance Scale From Baseline
Description: The Berg Balance Measure (Berg) was designed to test an elderly patient's level of balance. The test consists of 14 balance items that have been deemed safe for elderly patients to perform. The Berg is a task performance exam that takes about 15 to 20 minutes to complete. The test is scored while it is administered. Each of the independent items are scored on a five point ordinal scale where 0 indicates the patient's inability to perform the task and 4 represents independence; the individual points are then summed to achieve a total score (range 0 - 56). The higher the patient's score on the Berg the more independent the patient. The reported outcome is the change in the Berg between baseline and end of treatment.
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiveStep | Standard Treatment
Number analyzed (Participants) | 175 | 180
units on a scale | 5.96 (5.17) | 5.79 (5.22)

5. Secondary Outcome: Change in Dynamic Gait Index From Baseline
Description: The Dynamic Gait Index (DGI) is another instrument that was developed to assess the likelihood of falling in older adults and tests eight facets of gait. The DGI takes about 15 minutes and requires the following equipment: a Box (Shoebox); 2 Cones; Stairs; and a 20' walkway that is 15" wide. Each item is scored on a four-point ordinal scale, ranging from 0-3 where "0" indicates the lowest level of function and "3" the highest level of function, resulting in a total score of 0 to 24. The interpretation guidelines state that a score < 19/24 is predictive of falls in the elderly while as score of > 22/24 indicate safe walkers. The outcome reported is the change in the DGI between baseline and end-of-treatment.
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiveStep | Standard Treatment
Number analyzed (Participants) | 172 | 177
units on a scale | 3.26 (5.7) | 3.74 (3.37)

6. Secondary Outcome: Change in Activities-specific Balance Confidence From Baseline
Description: The Activity-specific Balance Confidence scale (ABC) is a patient self-report measure tthat measures the subject's self-assessed confidence in being able to perform 16 specific activities without losing their balance or becoming unsteady. For each task (i.e. walking around the house, sweeping the floor, walking outside on an icy sidewalk) the subject indicates their level of confidence in doing the activity without losing their balance. For items the subject does not normally perform, they are asked to try and imagine how confident they would feel if they had to do the activity. For subjects who normally use a walking aid to do the specific activity, they are asked to rate their confidence as if they were using these supports. Each item is rated 0-100 for each item. To obtain the final score, the ratings are averaged across the 16 items to produce an overall score from 0-100 with higher scores indicated greater balance confidence.
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiveStep | Standard Treatment
Number analyzed (Participants) | 177 | 168
units on a scale | 11.05 (16.08) | 12.05 (17.29)

ADVERSE EVENTS:
Groups:
- ActiveStep: Activestep Group
- Standard Treatment: Standard Treatment Group
Arm/Group | ActiveStep | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 13/245 | 6/245
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/245
Other Adverse Events (participants affected / at risk) | 0/245 | 0/245

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No